CLINICAL TRIAL: NCT01868906
Title: Positron Emission Tomography With Fluoro-misonidazole (PET-FMISO) in High Grade Gliomas: Assessment of Tumor Hypoxia and Effect of Spinal Cord Stimulation
Brief Title: FMISO-PET in Brain Tumors and SCS Effect
Acronym: FMISOPETSCS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Isotope (FMISO) production is no longer available in our country.
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Instituto Tecnologico Servicios Sanitarios, in MD Anderson Cancer Center, Madrid (Unknown); Instituto de Salud Carlos III (Other Government); Grupo de Investigación Clínica en Oncología Radioterapia (Other); Instituto Canario de Investigación del Cáncer (Other); RSbiomed (Unknown); Fundación DISA, Canary Islands, Spain (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, Radiation Oncologist, MD, PhD, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TC-FMISO-PET-06-1413; 2009-015852-11 (EudraCT Number); PI 06/1413, PI 12/02940 (Other Grant/Funding Number: Instituto de Salud Carlos III); TC-FMISO-PET-06-1413 (Other: Dr. Negrin University Hospital)
Record Dates: First submitted 2010-05-24; First posted 2013-06-05 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Malignant Glioma
Keywords: Anaplastic Astrocytoma; Brain Tumors; Cancer Imaging; Fluoromisonidazole; FMISO PET; Glioblastoma; High Grade Glioma; Hypoxia Modification; Positron Emission Tomography; Radiation-Sensitizing Agents; Spinal Cord Stimulation; Tumor Hypoxia Measurement
MeSH Terms: conditions — Glioma; Astrocytoma; Brain Neoplasms; Glioblastoma | interventions — fluoromisonidazole; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Spinal Cord Stimulation; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm-A: 18F-FMISO-PET without SCS (Other): One 18F-FMISO-PET study for assessment of tumor hypoxia before radiotherapy and Temozolomide, without spinal cord stimulation.
  Interventions: Drug: 18F-FMISO; Procedure: PET without SCS; Radiation: Radiotherapy; Drug: Temozolomide
- Arm-B: 18F-FMISO-PET without/with SCS (Other): Two 18F-FMISO-PET studies for assessment of tumor hypoxia before radiotherapy and Temozolomide: one "without" and one "with" spinal cord stimulation
  Interventions: Drug: 18F-FMISO; Procedure: PET without SCS; Device: SCS; Procedure: PET without/with SCS; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Drug: 18F-FMISO — 18F-FMISO-PET scanning, for tumor hypoxia assessment before radio-chemotherapy.
  Other Names: Fluoromisonidazole; FMISO
Procedure: PET without SCS — PET-scanning using 18F-fluoromisonidazole without SCS
  Other Names: Positron emission tomography scanning
Device: SCS — Electrical stimulation of spinal cord, minimally invasive neurosurgical technique used to treat refractory pain and ischemic syndromes.
  Other Names: Electrical Neurostimulation; Spinal Cord Stimulation
  Arms: Arm-B: 18F-FMISO-PET without/with SCS
Procedure: PET without/with SCS — Second PET-scanning using 18F-fluoromisonidazole: without/with SCS
  Other Names: Positron emission tomography scanning
  Arms: Arm-B: 18F-FMISO-PET without/with SCS
Radiation: Radiotherapy — Standard radiation therapy
  Other Names: Radiation therapy
Drug: Temozolomide — Standard treatment with concurrent and adjuvant Temozolomide.
  Other Names: Temodar; Temodal; Temcad

SUMMARY:
The aim of this study is to assess, with 18F-FMISO PET, hypoxia in high grade gliomas and changes by spinal cord stimulation in a subset of patients. Additionally, the potential correlation with pathological, imaging and clinical parameters will be analyzed.

DETAILED DESCRIPTION:
Tumour ischaemia-hypoxia decreases the efficacy of radio-chemotherapy. Polarographic probe (and some 18F-FMISO-PET) studies have demonstrated prognostic value. Additionally hypoxia modification may increase survival. However, in high grade gliomas (HGG) there are not well established methods to evaluate and modify tumor hypoxia. We have previously described how spinal cord stimulation (SCS) can modify oxygenation, blood flow and metabolism in malignant gliomas. The aim of this study is to assess with 18F-FMISO PET: hypoxia in HGG and changes by spinal cord stimulation in a subset of patients. Additionally, the potential correlation with pathological, imaging and clinical parameters will be analyzed.

18F-FMISO PET will be performed in 20 patients with diagnosis of HGG: after surgery/biopsy and before radical treatment with 3D radiotherapy and temozolomide. A subset of 10 patients undergo two studies with 18F- FMISO-PET (one with SCS "off" and one with SCS "on"). In these patients, SCS will be connected from 1 hour before to 1 hour after each radiotherapy session, and in the day-time during the days of adjuvant temozolomide.

18F-FMISO PET results will not be taking into account for patient management. Patients will be followed at least until the end of adjuvant temozolomide (6 months after the end of concurrent radiochemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed (first presentation or relapsed) high grade glioma (Grade III or Grade IV according WHO criteria) proposed for radical treatment with 3D radiotherapy and temozolomide.
* Patients 18-75 years old.
* Karnofsky >= 60% and ECOG =< 2.
* Signed informed consent.

Exclusion Criteria:

* Clinical or psychological contraindications to fly (if 18F-FMISO-PET is realized in Madrid) or to SCS-placement (only for this subset).
* Pregnant or breastfeeding women and women of fertile age who are not using a safe contraceptive method or do not intend to use one during the trial. Safe contraceptive methods are oral or parenteral contraceptive treatments or barrier methods: masculine or feminine condom, diaphragm and/or intrauterine device (IUD) or withdrawal over the course of the study.
* Serious co-existing or concurrent illness, including any of the following: uncontrolled or severe infection, heart, liver or kidney disease
* Lung thromboembolism.
* Another malignancy in the last 5 years other than basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patients with life expectancy <3 months.
* Patients with any of the following: creatinine > 2 mg/dl, neutrophils <1.5 * 10^9/L, platelets <100 * 10^9/L or hemoglobin <8.5 g/dL.
* Contraindications to receive radiotherapy or chemotherapy Clinical or psychological contraindications for placement of spinal cord stimulation devices (only for that specific subset of patients).
* Patients who are unable or unwilling to meet the protocol study.
* Patients who do not meet all the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06; Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Tumor hypoxia measurement using 18F-FMISO-PET (hypoxic volume and tumor/muscle ratio). Baseline measurement. | 18F-FMISO-PET between 1 and 3 weeks before the commencement of radio-chemotherapy
  Tumor hypoxia will be measured in 20 patients with HGG using 18F-FMISO-PET: after biopsy or surgery and before the commencement of radio-chemotherapy. It will be assessed the prevalence and extent of significant hypoxia in HGG.
Change from baseline tumor hypoxia using 18F-FMISO-PET (hypoxic volume and tumor/muscle ratio) during SCS. | 2nd 18F-FMISO-PET between 1 and 7 days after the 1st 18F-FMISO-PET
  A subset of 10 patients will undergo a second 18F-FMISO-PET study during spinal cord stimulation to evaluate changes by SCS between 1 and 7 days after the first 18F-FMISO-PET study (and before the commencement of radio-chemotherapy).

SECONDARY OUTCOMES:
Correlation between 18F-FMISO-PET values and pathological tumor parameters | Week 0 (at the commencement of radio-chemotherapy).
  To analyze the correlation of 18F-FMISO-PET with histological parameters and tumor expression of: CD31 (vascular density), VEGF (vascular endothelial growth factor) and VEGFR (angiogenesis), EGFR (epidermal growth factor receptor), Ki-67 (proliferation index) and hypoxic markers
Correlation with Karnofsky scale. | At 0, 2 and 9 months after the commencement of the radio-chemotherapy.
  To analyze the correlation with performance status using the Karnofsky scale.
Correlation with the ECOG (Eastern Cooperative Oncology Group) performance status scale | At 0, 2 and 9 months after the commencement of the radio-chemotherapy
  To analyze the correlation with performance status using the ECOG (WHO) scale.
Correlation with the Quality of Life Questionnaire QLQ-C30 (EORTC) | At 0, 2 and 9 months after the commencement of the radio-chemotherapy.
  To analyze the correlation with quality of life using the QLQ-C30 (EORTC) questionnaire.
Overall survival. | At 9 months after the commencement of the radio-chemotherapy.
  To analyze the correlation with overall survival.
Radiological response to treatment | 9 months after the commencement of radio-chemotherapy
  To analyze the correlation between 18F-FMISO-PET values and radiological response to treatment
Radiological location of tumor relapse or progression | 9 months after the commencement of radio-chemotherapy
  To analyze the correlation between 18F-FMISO-PET values and the radiological location of tumor relapse or progression

OTHER OUTCOMES:
Blood flow in carotid and middle cerebral arteries | Between 1 and 3 weeks before the commencement of radio-chemotherapy
  To analyze the correlation between 18F-FMISO-PET values and blood flow in carotid and middle cerebral arteries (assessed before the commencement of radio-chemotherapy) using Doppler measurements.
Facial and supraciliar infrared emission | Between 1 and 3 weeks before the commencement of radio-chemotherapy
  To analyze the correlation between 18F-FMISO-PET values and facial and supraciliar infrared emission (assessed by digital thermography)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Dr. Negrin University Hospital, Las Palmas; Bernardino Clavo, MD, PhD, Principal Investigator — Dr. Negrin University Hospital, Las Palmas; Francisco Robaina, MD, PhD, Principal Investigator — Dr. Negrin University Hospital, Las Palmas; Juan C Alonso, MD, PhD, Principal Investigator — Instituto Tecnologico Servicios Sanitarios, in MD Anderson Cancer Center, Madrid
Locations (2):
- Spain (2):
  - Dr. Negrin University Hospital, Las Palmas
  - Instituto Tecnologico Servicios Sanitarios, in MD Anderson Cancer Center, Madrid, Madrid

REFERENCES:
- [Background] Clavo B, Robaina F, Morera J, Ruiz-Egea E, Perez JL, Macias D, Carames MA, Catala L, Hernandez MA, Gunderoth M. Increase of brain tumor oxygenation during cervical spinal cord stimulation. Report of three cases. J Neurosurg. 2002 Jan;96(1 Suppl):94-100. doi: 10.3171/spi.2002.96.1.0094. PMID 11795721
- [Background] Clavo B, Robaina F, Catala L, Valcarcel B, Morera J, Carames MA, Ruiz-Egea E, Panero F, Lloret M, Hernandez MA. Increased locoregional blood flow in brain tumors after cervical spinal cord stimulation. J Neurosurg. 2003 Jun;98(6):1263-70. doi: 10.3171/jns.2003.98.6.1263. PMID 12816274
- [Background] Clavo B, Robaina F, Catala L, Perez JL, Lloret M, Carames MA, Morera J, Lopez L, Suarez G, Macias D, Rivero J, Hernandez MA. Effect of cervical spinal cord stimulation on regional blood flow and oxygenation in advanced head and neck tumours. Ann Oncol. 2004 May;15(5):802-7. doi: 10.1093/annonc/mdh189. PMID 15111351
- [Background] Clavo B, Robaina F, Montz R, Domper M, Carames MA, Morera J, Pinar B, Hernandez MA, Santullano V, Carreras JL. Modification of glucose metabolism in brain tumors by using cervical spinal cord stimulation. J Neurosurg. 2006 Apr;104(4):537-41. doi: 10.3171/jns.2006.104.4.537. PMID 16619657
- [Background] Robaina F, Clavo B, Catala L, Carames MA, Morera J. Blood flow increase by cervical spinal cord stimulation in middle cerebral and common carotid arteries. Neuromodulation. 2004 Jan;7(1):26-31. doi: 10.1111/j.1525-1403.2004.04003.x. PMID 22151123
- [Background] Clavo B, Robaina F, Montz R, Carames MA, Otermin E, Carreras JL. Effect of cervical spinal cord stimulation on cerebral glucose metabolism. Neurol Res. 2008 Jul;30(6):652-4. doi: 10.1179/174313208X305373. Epub 2008 May 29. PMID 18513465
- [Background] Clavo B, Robaina F, Montz R, Carames MA, Lloret M, Ponce P, Hernandez MA, Carreras JL. Modification of glucose metabolism in radiation-induced brain injury areas using cervical spinal cord stimulation. Acta Neurochir (Wien). 2009 Nov;151(11):1419-25. doi: 10.1007/s00701-009-0400-8. Epub 2009 Jun 5. PMID 19499176
- [Background] Clavo B, Robaina F, Valcarcel B, Catala L, Perez JL, Cabezon A, Jorge IJ, Fiuza D, Hernandez MA, Jover R, Carreras JL. Modification of loco-regional microenvironment in brain tumors by spinal cord stimulation. Implications for radio-chemotherapy. J Neurooncol. 2012 Jan;106(1):177-84. doi: 10.1007/s11060-011-0660-z. Epub 2011 Jul 12. PMID 21748490
- [Background] Overgaard J. Hypoxic radiosensitization: adored and ignored. J Clin Oncol. 2007 Sep 10;25(26):4066-74. doi: 10.1200/JCO.2007.12.7878. PMID 17827455
- [Background] Spence AM, Muzi M, Swanson KR, O'Sullivan F, Rockhill JK, Rajendran JG, Adamsen TC, Link JM, Swanson PE, Yagle KJ, Rostomily RC, Silbergeld DL, Krohn KA. Regional hypoxia in glioblastoma multiforme quantified with [18F]fluoromisonidazole positron emission tomography before radiotherapy: correlation with time to progression and survival. Clin Cancer Res. 2008 May 1;14(9):2623-30. doi: 10.1158/1078-0432.CCR-07-4995. PMID 18451225
- [Background] Clavo B, Robaina F, Jorge IJ, Cabrera R, Ruiz-Egea E, Szolna A, Otermin E, Llontop P, Carames MA, Santana-Rodriguez N, Sminia P. Spinal cord stimulation as adjuvant during chemotherapy and reirradiation treatment of recurrent high-grade gliomas. Integr Cancer Ther. 2014 Nov;13(6):513-9. doi: 10.1177/1534735414550037. Epub 2014 Sep 15. PMID 25228535
- [Background] Clavo B, Robaina F, Fiuza D, Ruiz A, Lloret M, Rey-Baltar D, Llontop P, Riveros A, Rivero J, Castaneda F, Quintero S, Santana-Rodriguez N. Predictive value of hypoxia in advanced head and neck cancer after treatment with hyperfractionated radio-chemotherapy and hypoxia modification. Clin Transl Oncol. 2017 Apr;19(4):419-424. doi: 10.1007/s12094-016-1541-x. Epub 2016 Aug 15. PMID 27527617